CLINICAL TRIAL: NCT06462976
Title: The Effect of Intraoperative Position and Mechanical Power on Postoperative Pulmonary Complications in Adult PNL(Percutaneous Nephrolithotomy) Patients
Brief Title: Postoperative Pulmonary Complications in Adult PNL Patients
Status: Recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gamze Talih, Principal Investigator, TC Erciyes University
Other Study IDs: 2024/99
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pulmonary Complication; Mechanical Power

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- supine: Which group the patients will be included in will be determined by the surgical team based on the location and number of stones. The patient's values will be recorded in that position.
  Interventions: Other: mechanical power calculation
- prone: Which group the patients will be included in will be determined by the surgical team based on the location and number of stones. The patient's values will be recorded in that position.
  Interventions: Other: mechanical power calculation

INTERVENTIONS:
Other: mechanical power calculation — Mechanical Power= 0.098×Minute ventilation× (peak pressure - 0.5 (plato pressure-PEEP)). These parameters are monitored on the monitor while the patient is mechanically ventilated and placed into the equation

SUMMARY:
The aim of this study is to investigate the effect of different surgical positions (supine/prone) on lung mechanical power (MP) and its relationship with postoperative pulmonary complications in patients planned to percutaneous nephrolithotomy (PNL) under general anesthesia.

DETAILED DESCRIPTION:
PNL is the preferred treatment method for kidney stones larger than 2 cm, multiple kidney stones and staghorn stones. With new developments in the field of medicine, PNL has become a minimally invasive method and is preferred to open surgery in the treatment of kidney stones. Alternative types of anesthesia and various patient positions have been described in PNL.

Mechanical power of ventilation (MP) is the amount of energy transferred from the mechanical ventilator to the respiratory system per unit time. Although this energy is primarily used to overcome airway resistance and respiratory system compliance, some of it acts directly on lung tissue, potentially causing ventilator-induced lung injury (VILI).

Mechanical power during ventilation estimates the energy delivered to the respiratory system by integrating inspiratory pressures, tidal volume and respiratory rate into a single value. It allows physicians to evaluate adjustments made to mechanical ventilation by calculating a single value. High mechanical power value is associated with a high incidence of postoperative pulmonary complications and mortality . In short, the energy distributed to the respiratory system consists of the static composite (PEEP), the dynamic composite (driving pressure and tidal volume) and the resistive composite (the pressure required for gas flow). Because energy is equal to the pressure that causes a change in volume. The equation is as follows: MP= 0.098 × respiratory rate × tidal volume × (PEEP + ½(plateau-peep)+ (peak-plateau)). These parameters are monitored on the monitor while the patient is mechanically ventilated and placed into the equation.

After general anesthesia, some postoperative pulmonary complications may be encountered. Exposure to high mechanical force in ventilated patients during surgery has been found to be associated with an increase in postoperative pulmonary complications and acute respiratory failure. This increases the length of hospital stay and mortality. In order to prevent ventilator-related lung damage, the mechanical ventilator must be adjusted to transfer the least amount of energy per unit time to the respiratory system for each patient.

Early recognition of postoperative pulmonary complications that are likely to occur after surgery is important for rapid initiation of treatment. Incentive spirometry (triflo) can be used to make a rapid assessment of the respiratory capacity of patients. An incentive spirometer is a device that measures the volume of air drawn into the lungs during inspiration. As you breathe through an incentive spirometer, a piston inside the device rises and measures the volume of inhaled air. 1 ball is considered as 600ml, 2 balls as 900ml, and 3 balls as 1200ml flow.]

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective percutaneous nephrolithotomy and agree to participate in the study.
* ASA 1-3 patient

Exclusion Criteria:

* Patients with acute and chronic hypoxemia (PaO2<65mmHg, SpO2<95 in room air)
* Patients with BMI>35
* Patients with obstructive sleep apnea syndrome
* Patients with ASA 4 and above
* Pregnant patients
* Pneumonia, COPD attack etc. before the operation. people with lung disease
* Unstable patients such as uncontrolled hypertension, decompensated heart
* Mentally retarded and uncooperative patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are aged 18-75 agree to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
mechanical power | 2 year
  mechanical power=0.098*minute ventilation *(Ppeak-0.5*(Pplato-PEEP)

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Talih, Kayseri, Kayseri, Turkey (Türkiye)